CLINICAL TRIAL: NCT05020665
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Entospletinib in Combination With Intensive Induction and Consolidation Chemotherapy in Adults With Newly Diagnosed Nucleophosmin 1-mutated Acute Myeloid Leukemia
Brief Title: Entospletinib Plus Intensive Induction/Consolidation Chemotherapy in Newly Diagnosed NPM1-mutated AML
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination was due to significant challenges associated with study enrollment in a genetic subset of fit participants in the front-line acute myeloid leukemia (AML) setting and other challenges associated with post-COVID impacts.
Sponsor: Kronos Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KB-ENTO-3001; 2021-000761-33 (EudraCT Number)
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Nucleophosmin 1-mutated Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Nucleophosmin 1-mutated Acute Myeloid Leukemia; Entospletinib; ENTO
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; Cytarabine; Anthracyclines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intensive Chemotherapy + Entospletinib (ENTO) (Experimental): Participants received intensive chemotherapy (cytarabine and anthracycline [daunorubicin or idarubicin]) in combination with entospletinib (ENTO).
  Interventions: Drug: Entospletinib; Drug: Cytarabine; Drug: Anthracycline
- Intensive Chemotherapy + Placebo (Placebo Comparator): Participants received intensive chemotherapy (cytarabine and anthracycline [daunorubicin or idarubicin]) in combination with the matching placebo.
  Interventions: Drug: Placebo; Drug: Cytarabine; Drug: Anthracycline

INTERVENTIONS:
Drug: Entospletinib — 400 mg, Orally as tablets
  Other Names: ENTO; GS-9973
  Arms: Intensive Chemotherapy + Entospletinib (ENTO)
Drug: Placebo — Orally as tablets
  Arms: Intensive Chemotherapy + Placebo
Drug: Cytarabine — Continuous infusion
Drug: Anthracycline — Either daunorubicin or idarubicin was administered via slow intravenous (IV) push

SUMMARY:
The primary objective of this study is to evaluate the efficacy of entospletinib (ENTO) compared to placebo when added to chemotherapy in previously untreated nucleophosmin-1 mutated (NPM1-m) acute myeloid leukemia (AML), as defined by the rate of molecularly defined measurable residual disease (MRD).

DETAILED DESCRIPTION:
This is a multi-center, international, double-blind, placebo-controlled study in previously untreated participants with acute myeloid leukemia (AML) harboring nucleophosmin-1 (NPM1) mutations. Upon fulfillment of all eligibility criteria, participants were randomized 1:1 to receive intensive chemotherapy in combination with either the spleen tyrosine kinase (SYK) inhibitor entospletinib (ENTO), or placebo. The study consisted of Screening, Induction, Consolidation, End-of-Treatment, and Long-term Follow-up phases.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 74 years with previously untreated de novo acute myeloid leukemia (AML), AML with myelodysplastic syndromes (MDS) features, or therapy-related AML, who were candidates for intensive induction therapy.
2. Nucleophosmin-1 (NPM1)-mutated disease documented in a local or the Sponsor's central testing facility.

   Note: Participants with local test results for nucleophosmin-1 mutated (NPM1-m) (and/or FMS-like tyrosine kinase 3 mutational status) may enroll, provided appropriate samples were sent to the Sponsor's central testing facility for NPM1-m companion diagnostic development.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0, 1, or 2.
4. Adequate hepatic and renal function defined as:

   1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times the upper limit of normal (ULN), except those with hepatic involvement by AML, as documented by either computed tomography (CT) or ultrasound, in whom levels of AST and ALT < 5 times ULN are acceptable; total bilirubin < 1.5 times ULN unless elevated due to Gilbert's Disease or hemolysis.
   2. Calculated creatinine clearance > 40 mL/min or serum creatinine < 1.5 times ULN.
5. Prothrombin time (PT), activated partial thromboplastin time (aPTT), and international normalized ratio (INR) ≤ 1.5 x ULN unless receiving therapeutic anticoagulation.
6. Left ventricular ejection fraction ≥ 45% confirmed by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan.

Exclusion Criteria:

1. Isolated myeloid sarcoma (ie, participants must had peripheral blood and/or bone marrow involvement by AML) or acute promyelocytic leukemia.
2. Concurrent FLT3 mutation (either tyrosine kinase domain or internal tandem duplication).
3. Known central nervous system (CNS) involvement with leukemia.
4. Was a candidate for more intensive treatment than specified in this protocol.
5. Either not a candidate for any anthracycline therapy or a candidate for induction therapy with a higher dose of daunorubicin (eg. 90 mg/m^2).
6. Was a candidate for daily doses of cytarabine > 100 mg/m^2 in Induction Cycle 1.
7. Active infection with hepatitis B, C, or uncontrolled human immunodeficiency virus (HIV).
8. Known active coronavirus disease 2019 (COVID-19) either symptomatic or asymptomatic, as determined by nasopharyngeal swab for severe acute respiratory syndrome (SARS) coronavirus 2 (SARS CoV-2) ribonucleic acid (RNA) or antigen.

   Note: Participants with a history of SARS-CoV-2 nasopharyngeal carriage (either with or without symptoms), who had subsequently tested negative on follow-up nasopharyngeal swab and were without signs or symptoms of COVID-19 might enroll. Participants who were fully vaccinated against SARS-CoV-2 might enroll.
9. Disseminated intravascular coagulation with active bleeding or signs of thrombosis.
10. History of prior allogeneic hematopoietic stem cell transplant or solid organ transplant.
11. Treatment with proton pump inhibitors (PPIs) from 7 days prior to enrollment until 48 hours after completion of entospletinib (ENTO) or placebo.

    Note: PPIs were likely to interfere with ENTO absorption, thus requiring a 7-day washout period prior to the initiation of study medication. For management of acute gastrointestinal bleeding during the study treatment period (such as that related to chemotherapy), short term concurrent use of PPIs was permitted for up to 10 consecutive days. If longer durations of PPI exposure were required, participants should discontinue study medication. Histamine (H2) receptor antagonists and antacids were allowed throughout the study treatment period.
12. Ongoing immunosuppressive therapy, including systemic chemotherapy for treatment of leukemia.

    Note: Participants may not receive AML-directed therapy prior to enrollment other than hydroxyurea or leukapheresis for acute management of hyperleukocytosis.
13. Clinical signs/symptoms of leukostasis that had failed therapy including hydroxyurea and/or leukapheresis of at least 3 days duration.
14. Clinically significant heart disease defined as:

    1. New York Heart Association Class 3 or 4 congestive heart failure,
    2. Acute myocardial infarction ≤ 6 months before enrollment,
    3. Symptomatic cardiac ischemia/unstable angina ≤ 3 months before enrollment,
    4. History of clinically significant arrhythmias (eg, ventricular tachycardia or fibrillation; Torsades de Pointe) including Mobitz type II 2nd degree or 3rd degree heart block without a permanent pacemaker in place.
15. Participants with a corrected congenital long measure between Q wave and T wave in the electrocardiogram (QT) interval (using the Fredericia formula, Fridericia correction of the QT measure [QTcF]) > 480 msec or Long QT Syndrome.
16. Evidence of ongoing, uncontrolled systemic bacterial, fungal, or viral infection at the time of study treatment initiation, including but not limited to persistent fever or positive cultures in the setting of appropriate antimicrobial therapy.
17. Unable to swallow tablets or concurrent disease affecting gastrointestinal function such as, malabsorption syndrome, gastric or small bowel resection, bariatric surgery, inflammatory bowel disease, or bowel obstruction.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (10):
  - City of Hope, Duarte, California
  - UCLA - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Indiana Blood & Marrow Transplantation, Indianapolis, Indiana
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mount Sinai Health System, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Hollings Cancer Center, Charleston, South Carolina
  - Bon Secours St. Francis Cancer Center, Greenville, South Carolina
  - Baylor University Medical Center, Dallas, Texas
- Brazil (9):
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba
  - Hospital Universitário Walter Cantídio, Fortaleza
  - Hospital Amaral Carvalho, Jaú
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia Hospital - Porto Alegre, Porto Alegre
  - Instituto Nacional de Câncer - Brazil, Rio de Janeiro
  - Hospital de Base - São José do Rio Preto, Rio Preto
  - A Beneficência Portuguesa de São Paulo - Unidade Mirante, São Paulo
  - Instituto Brasileiro de Controle do Câncer - São Camilo Oncologia - Unidade Mooca, São Paulo
- Canada (3):
  - Juravinski Hospital, Hamilton
  - Saskatchewan Cancer Agency, Saskatoon
  - Princess Margaret Cancer Centre, Toronto
- Czechia (3):
  - Fakultni Nemocnice Brno, Brno
  - Fakultní Nemocnice Hradec Králové, Hradec Králové
  - Fakultní Nemocnice Královské Vinohrady, Prague
- France (9):
  - Hôpital Côte De Nacre, Caen, Calvados
  - Centre Hosptitalier Universitaire d'Angers, Angers
  - Hôpital Claude Huriez, Lille
  - Hôpital l'Archet, Nice
  - Hôpital Saint-Antoine, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre de Lutte Contre le Cancer - Centre Henri-Becquerel, Rouen
- Germany (6):
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Helios St. Johannes Klinik, Duisburg
  - Marien Hospital Düsseldorf, Düsseldorf
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Münster, Münster
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Jósa András Oktatókórház, Nyíregyháza
  - Szent-Györgyi Albert Klinikai Központ, Szeged
- Israel (6):
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Hospital - Ramat HaHayal, Tel Aviv
- Italy (7):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania, Sicily
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico di Bari, Bari
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Ospedale Santa Maria delle Croci di Ravenna, Ravenna
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Nr im. Prof. Tadeusza Sokołowskiego, Szczecin
  - Uniwersyteckie Centrum Kliniczne WUM - Centralny Szpital Kliniczny, Warsaw
  - Instytut Hematologii I Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw
- South Korea (10):
  - Kyungpook National University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Catholic University of Korea Seoul Saint Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (10):
  - Hospital Germans Trias i Pujol, Badalona, Catalonia
  - Institut D'Investigacions Biomédiques August Pi I Sunyer, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Llàtzer, Palma de Mallorca
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 5 countries including the Czechia, France, Republic of Korea, Spain, and the United States from 24 November 2021 to 30 March 2023.
Pre-assignment Details: In this study participants were randomized 1:1 to receive intensive chemotherapy in combination with either the spleen tyrosine kinase inhibitor, entospletinib (ENTO), or placebo. Randomization was stratified by age (< 60 vs ≥ 60 years) and anthracycline administered during induction (daunorubicin vs idarubicin). In November 2022, the Sponsor decided to terminate this study prior to full enrollment.
Groups:
- ENTO: Participants received ENTO twice daily (BID), along with intensive chemotherapy (cytarabine and anthracycline) by continuous intravenous (IV) infusion (cytarabine) or slow IV push (anthracycline)
- Placebo: Participants received placebo BID, along with intensive chemotherapy (cytarabine and anthracycline) by continuous intravenous (IV) infusion (cytarabine) or slow IV push (anthracycline)
Period: Overall Study
Arm/Group | ENTO | Placebo
Started | 8 | 7
Completed | 0 | 0
Not Completed | 8 | 7
Not completed — Study terminated by Sponsor | 5 | 4
Not completed — Death | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Reason not specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ENTO | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (9.41) | 54.6 (16.11) | 55.7 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Measurable Residual Disease (MRD) Negative Complete Response (CR) Rate
Description: MRD negative CR requires CR as defined by the European Leukemia Network (ELN) 2017 criteria (with minor modification for neutrophil and platelet count thresholds as defined by International Working Group [IWG]) as assessed by study site investigators, and MRD negativity (<0.01%) in bone marrow as measured by a molecular nucleophosmin-1 mutated (NPM1-m) assay (eg, next generation sequencing) in a central laboratory upon recovery of peripheral blood counts following completion of 2 cycles of chemotherapy, no later than Day 42 of Cycle 2.
Time Frame: Cycle 1 Day 1, up to Day 42 of chemotherapy cycle 2 (Cycle length = 42 days)
Population: Data not collected as the study was terminated early.
Groups:
- ENTO: Participants received ENTO BID, along with intensive chemotherapy (cytarabine and anthracycline) by continuous IV infusion (cytarabine) or slow IV push (anthracycline).
- Placebo: Participants received placebo, BID, along with intensive chemotherapy (cytarabine and anthracycline) by continuous IV infusion (cytarabine) or slow IV push (anthracycline).
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the time from randomization to the earliest occurrence of induction treatment failure, relapse from CR, or death from any cause. Induction treatment failure is failure to achieve morphological CR after completion of the last cycle of induction chemotherapy (no later than Day 42 of the last cycle of induction).
Time Frame: Cycle 1 Day 1, up to Day 42 of chemotherapy cycle 2 (Cycle length = 42 days)
Population: Data not collected as the study was terminated early.
Groups:
- ENTO: Participants received ENTO, BID, along with intensive chemotherapy (cytarabine and anthracycline) by continuous IV infusion (cytarabine) or slow IV push (anthracycline).
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS is defined as the time from CR until relapse or death from any cause as assessed by study site investigators.
Time Frame: Cycle 1 Day 1, up to Day 42 of chemotherapy cycle 2 (Cycle length = 42 days)
Population: Data not collected as the study was terminated early.
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until death from any cause.
Time Frame: Cycle 1 Day 1, up to Day 42 of chemotherapy cycle 2 (Cycle length = 42 days)
Population: Data not collected as the study was terminated early.
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participant With Complete Response (CR) After 2 Cycles of Chemotherapy
Description: CR as defined by ELN 2017 criteria (with minor modification for neutrophil and platelet count thresholds as defined by IWG) as assessed by study site investigators.
Time Frame: Cycle 1 Day 1, up to Day 42 of chemotherapy cycle 2 (Cycle length = 42 days)
Population: Intent-to-Treat (ITT) Analysis Set: All participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 8 | 7
Participants | 5 | 5

6. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is any untoward medical occurrence in a clinical study participant, beginning or worsening from Cycle 1, Day 1 through 30 days following study treatment completion, temporarily associated with the use of treatment, whether or not considered related to the study treatment. TEAEs were recorded according to the most current version of the Medical Dictionary for Regulatory Activities (MedDRA).
  Clinically significant changes in safety laboratory assessments, electrocardiograms, echocardiogram / multi-gated acquisition scans and Eastern Cooperative Oncology Group performance status findings, as assessed by the Investigator, were recorded as TEAEs.
Time Frame: Cycle 1 Day 1 to 30 days following study treatment completion, (Cycle length = 42 days) maximum up to 198 days
Population: Safety Analysis Set: All participants randomized who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- ENTO: Participants received ENTO, BID along with intensive chemotherapy (cytarabine and anthracycline) by continuous IV infusion (cytarabine) or slow IV push (anthracycline).
Arm/Group | ENTO | Placebo
Number analyzed (Participants) | 8 | 7
Participants | 8 | 7

ADVERSE EVENTS:
Time Frame: Serious adverse events and deaths were collected from signing informed consent through 30 days after treatment completion, up to 212 days. Other adverse events were collected from Day 1 of Cycle 1 through 30 days after treatment completion, up to 198 days.
Description: A TEAE is any untoward medical occurrence in a clinical study participant, beginning or worsening from Cycle 1, Day 1 through 30 days following study treatment completion, temporarily associated with the use of treatment, whether or not considered related to the study treatment. TEAEs were recorded according to the most current version of the Medical Dictionary for Regulatory Activities (MedDRA).
Arm/Group | ENTO | Placebo
All-Cause Mortality (participants affected / at risk) | 3/8 | 1/7
Serious Adverse Events (participants affected / at risk) | 8/8 | 2/7
Other Adverse Events (participants affected / at risk) | 7/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENTO (N=8) | Placebo (N=7)
Klebsiella bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENTO (N=8) | Placebo (N=7)
Nausea (Gastrointestinal disorders) | 4 (7) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (5) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (4) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (29) | 3 (34)
Anaemia (Blood and lymphatic system disorders) | 3 (36) | 3 (25)
Neutropenia (Blood and lymphatic system disorders) | 2 (19) | 3 (20)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (16)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (4)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 1 (2)
Chills (General disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Deformity (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (4)
Pain (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 2 (4) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (12) | 3 (8)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (15) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (4)
Amylase increased (Investigations) | 1 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 1 (2)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (4)
Gamma-glutamyltransferase increased (Investigations) | 1 (4) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (3)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Cytarabine syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Renal cyst (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination was due to significant unforeseen challenges associated with global enrollment of participants with genetically-defined, newly diagnosed, AML who are candidates for intensive induction therapy and other challenges associated with post-COVID impacts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT05020665/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT05020665/SAP_001.pdf